CLINICAL TRIAL: NCT01545609
Title: A Text Message Support System for Effective Continuation of a Birth Control Method in Female Adolescents: 'BC 2U'
Brief Title: A Trial Assessing the Effectiveness of Text Messages in Improving Continuation of Birth Control
Acronym: BC 2U
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 11-1385; HS#: 11-01558
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Initiation of a Birth Control Method
Keywords: Text messaging; birth control; adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text messaging (Experimental): Text messaging
  Interventions: Other: Text messaging
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Other: Text messaging — Text messages to cell phone with education messages about the specific birth control they are using
  Arms: Text messaging

SUMMARY:
This study is a randomized controlled trial assessing the effectiveness in a series of educational text messages in improving continuation of a birth control method in comparison to the 'standard counseling', when girls initiate a new method of birth control. Girls aged 15-19 year olds who are attending for a reproductive health visit and who own a working cell phone will be approached and asked if they would like to participate. Following completion of a baseline questionnaire and consultation for initiation of a new birth control method they will be randomized to receive either the intervention or standard counseling.

If randomized to the intervention they will receive 3 messages per week for the initial 3 weeks, 2 messages per week for the following 5 weeks and then one message per week thereafter. Messages will be tailored to the birth control method the participant has initiated. At 4 months all participants will be contacted via telephone and asked to complete a questionnaire regarding continuation of use.

DETAILED DESCRIPTION:
Hypothesis. A personalized text messaging program providing trustworthy, reliable information and support to female adolescents initiating a birth control method, will improve adherence and correct use of the method and so reduce unwanted pregnancies.

Methods. Female adolescents aged 15-19 year olds attending Mount Sinai Adolescent Health Center (MSAHC) for initiating a birth control method will be asked if they are interested in participating in the trial.

The Intervention Group. Upon initiation of a birth control method patients will be signed up to the text messaging platform. Via this program they will receive personalized messages regarding their chosen method of birth control. Participants will receive 3 messages during the initial 3 weeks, 2 messages per week in weeks 4-8 and then one message a week thereafter for a period of 12 months. They will be signed up for reminders to take/change their method (as appropriate) and have access to a Healthcare Provider to ask questions via text message that they may have regarding their method. Participants will be reminded (via text message) to attend the clinic for a birth control refill (if necessary) at 3, 6, 9 and 12 months.

The Control Group. Participants randomized in to the control group will have standard care. This is the usual counseling by the Health Care Provider or Health Educator. Patients in the intervention arm will also receive this standard care.

ELIGIBILITY:
Inclusion Criteria:

* female
* Aged 15-19 years old
* English speaking
* owner of a working cell phone
* patient must be wanting to start a birth control method and not have been on a method for preceding 3 months
* no contra indications to initiating a birth control method

Exclusion Criteria:

* male
* younger than 15 years old, older than 19 years old
* already on a birth control method
* Not English speaking
* No working cell phone in possession

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Continuation of a birth control method | at 4 months
  Birth control continuation will be assessed at 4 months by direct asking of the participant to see if participant has attended for a refill of her birth control method.

SECONDARY OUTCOMES:
Change in birth control method being used. | at 4 months
  whether subjects continue with the initial method of birth control or discontinue a method at the 4 months.
Pregnancy | at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Francis, MD, Principal Investigator — Mount Sinai Adolescent Health Center
Locations (1):
- Mount Sinai Adolescent Health Center, New York, New York, United States

REFERENCES:
- [Background] Gilliam M, Knight S, McCarthy M Jr. Success with oral contraceptives: a pilot study. Contraception. 2004 May;69(5):413-8. doi: 10.1016/j.contraception.2003.12.006. PMID 15105065
- [Background] Woods JL, Shew ML, Tu W, Ofner S, Ott MA, Fortenberry JD. Patterns of oral contraceptive pill-taking and condom use among adolescent contraceptive pill users. J Adolesc Health. 2006 Sep;39(3):381-7. doi: 10.1016/j.jadohealth.2005.12.014. Epub 2006 Jul 10. PMID 16919800
- [Background] Moos MK, Bartholomew NE, Lohr KN. Counseling in the clinical setting to prevent unintended pregnancy: an evidence-based research agenda. Contraception. 2003 Feb;67(2):115-32. doi: 10.1016/s0010-7824(02)00472-9. PMID 12586322
- [Background] Bruckner H, Martin A, Bearman PS. Ambivalence and pregnancy: adolescents' attitudes, contraceptive use and pregnancy. Perspect Sex Reprod Health. 2004 Nov-Dec;36(6):248-57. doi: 10.1363/psrh.36.248.04. PMID 15687083
- [Background] Langston AM, Rosario L, Westhoff CL. Structured contraceptive counseling--a randomized controlled trial. Patient Educ Couns. 2010 Dec;81(3):362-7. doi: 10.1016/j.pec.2010.08.006. PMID 20869187
- [Background] Speizer IS, Santelli JS, Afable-Munsuz A, Kendall C. Measuring factors underlying intendedness of women's first and later pregnancies. Perspect Sex Reprod Health. 2004 Sep-Oct;36(5):198-205. doi: 10.1363/psrh.36.198.04. PMID 15519962
- [Background] Kavanaugh ML, Schwarz EB. Prospective assessment of pregnancy intentions using a single- versus a multi-item measure. Perspect Sex Reprod Health. 2009 Dec;41(4):238-43. doi: 10.1363/4123809. PMID 20444179
- [Background] Santelli J, Rochat R, Hatfield-Timajchy K, Gilbert BC, Curtis K, Cabral R, Hirsch JS, Schieve L; Unintended Pregnancy Working Group. The measurement and meaning of unintended pregnancy. Perspect Sex Reprod Health. 2003 Mar-Apr;35(2):94-101. doi: 10.1363/3509403. No abstract available. PMID 12729139
- [Background] Zabin LS, Astone NM, Emerson MR. Do adolescents want babies? The relationship between attitudes and behavior. J Res Adolesc. 1993;3(1):67-86. doi: 10.1207/s15327795jra0301_4. PMID 12318551
- [Background] Cowley C, Farley T. Adolescent girls' attitudes toward pregnancy: the importance of asking what the boyfriend wants. J Fam Pract. 2001 Jul;50(7):603-7. PMID 11485709
- [Background] Miller BC. Family influences on adolescent sexual and contraceptive behavior. J Sex Res. 2002 Feb;39(1):22-6. doi: 10.1080/00224490209552115. PMID 12476252
- [Background] Gold J, Lim MS, Hellard ME, Hocking JS, Keogh L. What's in a message? Delivering sexual health promotion to young people in Australia via text messaging. BMC Public Health. 2010 Dec 29;10:792. doi: 10.1186/1471-2458-10-792. PMID 21190584
- [Background] Adams BN, McAnarney ER, Panzarine S, Tuttle JI. Successful contraceptive behavior among adolescent mothers: are there predictors? J Adolesc Health Care. 1990 Jul;11(4):319-25. doi: 10.1016/0197-0070(90)90042-z. PMID 2365606
- [Background] Barnet B, Liu J, DeVoe M, Duggan AK, Gold MA, Pecukonis E. Motivational intervention to reduce rapid subsequent births to adolescent mothers: a community-based randomized trial. Ann Fam Med. 2009 Sep-Oct;7(5):436-45. doi: 10.1370/afm.1014. PMID 19752472
- [Background] Hall KS, Castano PM, Stone PW, Westhoff C. Measuring oral contraceptive knowledge: a review of research findings and limitations. Patient Educ Couns. 2010 Dec;81(3):388-94. doi: 10.1016/j.pec.2010.10.016. Epub 2010 Nov 16. PMID 21084170
- [Background] Jaccard J, Helbig DW, Wan CK, Gutman MA, Kritz-Silverstein DC. The prediction of accurate contraceptive use from attitudes and knowledge. Health Educ Q. 1996 Feb;23(1):17-33. doi: 10.1177/109019819602300102. PMID 8822399
- [Background] Jones RK, Kooistra K. Abortion incidence and access to services in the United States, 2008. Perspect Sex Reprod Health. 2011 Mar;43(1):41-50. doi: 10.1363/4304111. Epub 2011 Jan 10. PMID 21388504
- [Background] Lim MS, Hocking JS, Aitken CK, Fairley CK, Jordan L, Lewis JA, Hellard ME. Impact of text and email messaging on the sexual health of young people: a randomised controlled trial. J Epidemiol Community Health. 2012 Jan;66(1):69-74. doi: 10.1136/jech.2009.100396. Epub 2011 Mar 17. PMID 21415232
- [Background] U.S Teenage Pregnancies, Births, Abortions: National and State Trends and trends by Race and Ethnicity. Guttmacher Institute. January 2010.
- [Background] Pesa JA, Mathews J. The relationship between barriers to birth control use and actual birth control use among Mexican-American adolescents. Adolescence. 2000 Winter;35(140):695-707. PMID 11214208
- [Background] Lopez LM, Tolley EE, Grimes DA, Chen-Mok M. Theory-based interventions for contraception. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD007249. doi: 10.1002/14651858.CD007249.pub3. PMID 21412901
- [Background] Santelli JS, Lindberg LD, Finer LB, Singh S. Explaining recent declines in adolescent pregnancy in the United States: the contribution of abstinence and improved contraceptive use. Am J Public Health. 2007 Jan;97(1):150-6. doi: 10.2105/AJPH.2006.089169. Epub 2006 Nov 30. PMID 17138906
- [Background] Canto De Cetina TE, Canto P, Ordonez Luna M. Effect of counseling to improve compliance in Mexican women receiving depot-medroxyprogesterone acetate. Contraception. 2001 Mar;63(3):143-6. doi: 10.1016/s0010-7824(01)00181-0. PMID 11368986
- [Background] Jones RK, Kost K, Singh S, Henshaw SK, Finer LB. Trends in abortion in the United States. Clin Obstet Gynecol. 2009 Jun;52(2):119-29. doi: 10.1097/GRF.0b013e3181a2af8f. PMID 19407518
- [Background] Rose SB, Lawton BA, Brown SA. Uptake and adherence to long-acting reversible contraception post-abortion. Contraception. 2010 Oct;82(4):345-53. doi: 10.1016/j.contraception.2010.04.021. Epub 2010 May 26. PMID 20851228